CLINICAL TRIAL: NCT04457817
Title: CRI and Continuous Assessment of Hemodynamic Compensation to Guide Fluid and Pressor Management in Severely Ill Patients With COVID-19
Brief Title: Compensatory Reserve Index (CRI) for Management of COVID-19
Status: Terminated | Type: Observational
Why Stopped: Lack of feasibility
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1406
Record Dates: First submitted 2020-06-24; First posted 2020-07-07 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: COVID
Keywords: CRI; Compensatory Reserve Index; COVID-19; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CRI Monitoring/Management: These patients are COVID-19 positive; ages > 18 and < 70 years old; require > 2 liters of oxygen by nasal cannula to maintain SpO2 > 90%; are admitted to the sixth floor at University Hospital, on one of two designated Hospitalist services (approximately 16 COVID-19 positive patients/service). Patients in the study cohort will also be monitored with a CipherOx CR T1 tablet in a continuous manner to determine if maintaining CRI vales between 0.9-0.7 will: 1) help guide IV fluid (e.g. crystalloid, colloids, blood products) and medication therapy (e.g. diuretics); 2) allows earlier identification of patients who are poorly compensating and will require ICU level care; 3) reduces AKI and/or need for CRRT; and 4) improves clinical outcomes.
  Interventions: Device: CRI

INTERVENTIONS:
Device: CRI — Monitoring via CRI

SUMMARY:
The FDA has approved the CipherOx CRI T1 Tablet for use in subjects aged 19-36, and that this study aims to evaluate the device in subjects aged outside of this range and is being used off label.

The FDA determined the Cipher OX CRI T1 Tablet to be a class II device in 2016, and additional research has been done since the FDA determination to further support the use of the device outside of its current labeling.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will be those who are:

* COVID-19 positive;
* Ages > 18 and < 70 years old;
* Require > 2 liters of oxygen by nasal cannula to maintain SpO2 > 90%;
* Are admitted to the sixth floor at University Hospital, on one of two designated Hospitalist services (approximately 16 COVID-19 positive patients/service).

Exclusion Criteria:

* COVID-19 negative
* Age <18 or >70 years
* On <2 liters oxygen via nasal canula
* Pregnant
* Incarcerated
* DNR/DNI
* Decisionally Challenged

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 positive patients, Eligibility described above.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Volume of IV fluid infused | 1 year
  Volume of IV fluid infused during treatment
Quantity of Blood pressure medication administered | 1 year
  Amount of blood pressure medication utilized during treatment
Resuscitation status | 1 year
  Categorical determination of resuscitation status as over- or under- resuscitated
FiO2 needs | 1 year
  FiO2 levels administered
Days on Oxygen | 1 year
  Days spent on oxygen
Number of participants with hospital acquired pneumonia | 1 year
  Number of participants with hospital acquired pneumonia
Number of Patients with Acute Kidney Injury (AKI) | 1 year
  Number of patients who acquire an acute kidney injury
Number of patients with hemodynamic collapse | 1 year
  Number of patients who experience hemodynamic collapse defined as drop in systolic blood pressure below 80mm Hg
mortality | 1 year
  Number of patients who experience mortality

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Moulton, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Background] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: Guidelines on the Management of Critically Ill Adults with Coronavirus Disease 2019 (COVID-19). Crit Care Med. 2020 Jun;48(6):e440-e469. doi: 10.1097/CCM.0000000000004363. PMID 32224769
- [Background] Convertino VA, Moulton SL, Grudic GZ, Rickards CA, Hinojosa-Laborde C, Gerhardt RT, Blackbourne LH, Ryan KL. Use of advanced machine-learning techniques for noninvasive monitoring of hemorrhage. J Trauma. 2011 Jul;71(1 Suppl):S25-32. doi: 10.1097/TA.0b013e3182211601. PMID 21795890
- [Background] Moulton SL, Mulligan J, Grudic GZ, Convertino VA. Running on empty? The compensatory reserve index. J Trauma Acute Care Surg. 2013 Dec;75(6):1053-9. doi: 10.1097/TA.0b013e3182aa811a. PMID 24256681
- [Background] Convertino VA, Schiller AM. Measuring the compensatory reserve to identify shock. J Trauma Acute Care Surg. 2017 Jun;82(6S Suppl 1):S57-S65. doi: 10.1097/TA.0000000000001430. No abstract available. PMID 28333834
- [Background] Janak JC, Howard JT, Goei KA, Weber R, Muniz GW, Hinojosa-Laborde C, Convertino VA. Predictors of the Onset of Hemodynamic Decompensation During Progressive Central Hypovolemia: Comparison of the Peripheral Perfusion Index, Pulse Pressure Variability, and Compensatory Reserve Index. Shock. 2015 Dec;44(6):548-53. doi: 10.1097/SHK.0000000000000480. PMID 26529655
- [Background] Poh PY, Carter R 3rd, Hinojosa-Laborde C, Mulligan J, Grudic GZ, Convertino VA. Respiratory pump contributes to increased physiological reserve for compensation during simulated haemorrhage. Exp Physiol. 2014 Oct;99(10):1421-6. doi: 10.1113/expphysiol.2014.081208. Epub 2014 Jul 11. PMID 25016024
- [Background] Van Sickle C, Schafer K, Mulligan J, Grudic GZ, Moulton SL, Convertino VA. A sensitive shock index for real-time patient assessment during simulated hemorrhage. Aviat Space Environ Med. 2013 Sep;84(9):907-12. doi: 10.3357/asem.3606.2013. PMID 24024301
- [Background] Carter R 3rd, Hinojosa-Laborde C, Convertino VA. Variability in integration of mechanisms associated with high tolerance to progressive reductions in central blood volume: the compensatory reserve. Physiol Rep. 2016 Feb;4(4):e12705. doi: 10.14814/phy2.12705. PMID 26884477
- [Background] Hinojosa-Laborde C, Howard JT, Mulligan J, Grudic GZ, Convertino VA. Comparison of compensatory reserve during lower-body negative pressure and hemorrhage in nonhuman primates. Am J Physiol Regul Integr Comp Physiol. 2016 Jun 1;310(11):R1154-9. doi: 10.1152/ajpregu.00304.2015. Epub 2016 Mar 30. PMID 27030667
- [Background] Stewart CL, Mulligan J, Grudic GZ, Convertino VA, Moulton SL. Detection of low-volume blood loss: compensatory reserve versus traditional vital signs. J Trauma Acute Care Surg. 2014 Dec;77(6):892-7; discussion 897-8. doi: 10.1097/TA.0000000000000423. PMID 25423536
- [Background] Nadler R, Convertino VA, Gendler S, Lending G, Lipsky AM, Cardin S, Lowenthal A, Glassberg E. The value of noninvasive measurement of the compensatory reserve index in monitoring and triage of patients experiencing minimal blood loss. Shock. 2014 Aug;42(2):93-8. doi: 10.1097/SHK.0000000000000178. PMID 24667628
- [Background] Convertino VA, Howard JT, Hinojosa-Laborde C, Cardin S, Batchelder P, Mulligan J, Grudic GZ, Moulton SL, MacLeod DB. Individual-Specific, Beat-to-beat Trending of Significant Human Blood Loss: The Compensatory Reserve. Shock. 2015 Aug;44 Suppl 1:27-32. doi: 10.1097/SHK.0000000000000323. PMID 25565640
- [Background] Stewart CL, Mulligan J, Grudic GZ, Talley ME, Jurkovich GJ, Moulton SL. The Compensatory Reserve Index Following Injury: Results of a Prospective Clinical Trial. Shock. 2016 Sep;46(3 Suppl 1):61-7. doi: 10.1097/SHK.0000000000000647. PMID 27172155
- [Background] Johnson MC, Alarhayem A, Convertino V, Carter R 3rd, Chung K, Stewart R, Myers J, Dent D, Liao L, Cestero R, Nicholson S, Muir M, Schwacha M, Wampler D, DeRosa M, Eastridge B. Compensatory Reserve Index: Performance of A Novel Monitoring Technology to Identify the Bleeding Trauma Patient. Shock. 2018 Mar;49(3):295-300. doi: 10.1097/SHK.0000000000000959. PMID 28767544
- [Background] Johnson MC, Alarhayem A, Convertino V, Carter R 3rd, Chung K, Stewart R, Myers J, Dent D, Liao L, Cestero R, Nicholson S, Muir M, Schwaca M, Wampler D, DeRosa M, Eastridge BJ. Comparison of compensatory reserve and arterial lactate as markers of shock and resuscitation. J Trauma Acute Care Surg. 2017 Oct;83(4):603-608. doi: 10.1097/TA.0000000000001595. PMID 28930955
- [Background] Choi YM, Leopold D, Campbell K, Mulligan J, Grudic GZ, Moulton SL. Noninvasive monitoring of physiologic compromise in acute appendicitis: New insight into an old disease. J Pediatr Surg. 2018 Feb;53(2):241-246. doi: 10.1016/j.jpedsurg.2017.11.013. Epub 2017 Nov 13. PMID 29217323
- [Background] Benov A, Brand A, Rozenblat T, Antebi B, Ben-Ari A, Amir-Keret R, Nadler R, Chen J, Chung KK, Convertino VA, Paran H. Evaluation of sepsis using compensatory reserve measurement: A prospective clinical trial. J Trauma Acute Care Surg. 2020 Aug;89(2S Suppl 2):S153-S160. doi: 10.1097/TA.0000000000002648. PMID 32118823
- [Background] Gagnon D, Schlader ZJ, Adams A, Rivas E, Mulligan J, Grudic GZ, Convertino VA, Howard JT, Crandall CG. The Effect of Passive Heat Stress and Exercise-Induced Dehydration on the Compensatory Reserve During Simulated Hemorrhage. Shock. 2016 Sep;46(3 Suppl 1):74-82. doi: 10.1097/SHK.0000000000000653. PMID 27183303
- [Background] Ehrmann DE, Leopold DK, Phillips R, Shahi N, Campbell K, Ross M, Zablah JE, Moulton SL, Morgan G, Kim JS. The Compensatory Reserve Index Responds to Acute Hemodynamic Changes in Patients with Congenital Heart Disease: A Proof of Concept Study. Pediatr Cardiol. 2020 Aug;41(6):1190-1198. doi: 10.1007/s00246-020-02374-3. Epub 2020 May 30. PMID 32474738
- [Background] Stewart CL, Mulligan J, Grudic GZ, Pyle L, Moulton SL. A noninvasive computational method for fluid resuscitation monitoring in pediatric burns: a preliminary report. J Burn Care Res. 2015 Jan-Feb;36(1):145-50. doi: 10.1097/BCR.0000000000000178. PMID 25383980
- [Background] Stewart CL, Nawn CD, Mulligan J, Grudic G, Moulton SL, Convertino VA. Compensatory Reserve for Early and Accurate Prediction of Hemodynamic Compromise: Case Studies for Clinical Utility in Acute Care and Physical Performance. J Spec Oper Med. 2016 Spring;16(1):6-13. PMID 27045488
- [Background] Leopold DK, Phillips RC, Shahi N, Gien J, Marwan AI, Kinsella JP, Mulligan J, Liechty KW, Moulton SL. Low postnatal CRI values are associated with the need for ECMO in newborns with CDH. J Pediatr Surg. 2020 Jan;55(1):39-44. doi: 10.1016/j.jpedsurg.2019.09.050. Epub 2019 Oct 25. PMID 31679772
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] Alexander PMA, DiOrio M, Andren K, Gauvreau K, Mistry KP, Mathieu D, Wright J, Allan CK, Nathan M, Mayer JE Jr, Thiagarajan RR, Bergersen L. Accurate Prediction of Congenital Heart Surgical Length of Stay Incorporating a Procedure-Based Categorical Variable. Pediatr Crit Care Med. 2018 Oct;19(10):949-956. doi: 10.1097/PCC.0000000000001668. PMID 30052551
- [Background] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Convertino VA, Wampler MR, Johnson M, Alarhayem A, Le TD, Nicholson S, Myers JG, Chung KK, Struck KR, Cuenca C, Eastridge BJ. Validating clinical threshold values for a dashboard view of the compensatory reserve measurement for hemorrhage detection. J Trauma Acute Care Surg. 2020 Aug;89(2S Suppl 2):S169-S174. doi: 10.1097/TA.0000000000002586. PMID 31972755
- [Background] Silversides JA, Major E, Ferguson AJ, Mann EE, McAuley DF, Marshall JC, Blackwood B, Fan E. Conservative fluid management or deresuscitation for patients with sepsis or acute respiratory distress syndrome following the resuscitation phase of critical illness: a systematic review and meta-analysis. Intensive Care Med. 2017 Feb;43(2):155-170. doi: 10.1007/s00134-016-4573-3. Epub 2016 Oct 12. PMID 27734109
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Erickson SE, Martin GS, Davis JL, Matthay MA, Eisner MD; NIH NHLBI ARDS Network. Recent trends in acute lung injury mortality: 1996-2005. Crit Care Med. 2009 May;37(5):1574-9. doi: 10.1097/CCM.0b013e31819fefdf. PMID 19325464